CLINICAL TRIAL: NCT02023424
Title: An Open Label, Exploratory Study to Investigate the Treatment Effect og Glatiramer Acetate (Copaxone ®) on Girls Woth Rett Syndrome
Brief Title: An Open Label, Exploratory Study to Investigate the Treatment Effect of Glatiramer Acetate on Girls Woth Rett Syndrome
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof. Bruria Ben-Zeev MD, Head of pediatric neurology unit and Israeli Rett Cener, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-12-9855-BBZ-CTIL
Record Dates: First submitted 2013-12-23; First posted 2013-12-30 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-02

CONDITIONS: Rett Syndrome
Keywords: BDNF; GLATIRAMER ACETATE; RETT SYNDROME; COPAXONE; Bruria Ben-Zeev
MeSH Terms: conditions — Rett Syndrome | interventions — Glatiramer Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Copaxone (Experimental): Glatiramer Acetate (Copaxone® , Teva Pharmaceutical Industries Ltd.) 20 mg daily or in an interval determined in the Dose Setting period. Administration will be subcutaneous to various areas on the body: back of the upper arms (2 areas), front and outside of thighs (2 areas), upper buttocks/rear hips (2 areas), and stomach (the abdomen).
  Interventions: Drug: Glatiramer Acetate (Copaxone®)

INTERVENTIONS:
Drug: Glatiramer Acetate (Copaxone®) — GA is a potent inducer of Th2-cells and modulates these immune cells to secrete high levels of neurotrophic factors, particularly BDNF. The induced cells cross the blood brain barrier (BBB), accumulate in the CNS and express BDNF and other regulatory substances in situ.

SUMMARY:
Primary Objective: To test the hypothesis that 6 months treatment with glatiramer acetate (GA) decreases epileptiform activity in young girls with Rett syndrome.

Primary Safety Objective:To evaluate the safety and tolerability of 6 months treatment with GA in these patients.

Secondary Objectives:

1. To test the hypothesis that 6 months treatment with glatiramer acetate (GA) improves respiratory dysfunction.
2. To evaluate the effect of GA treatment on general behaviour communication, hand stereotyping, feeding, sleep and other autonomic symptoms: gastrointestinal and cardiac.
3. To assess the effect of GA treatment on bodily development.

Primary Endpoint:Improvement of epileptiform activity as recorded in a 24-hours EEG.

Primary Safety Endpoint:Frequency and severity of treatment-related AEs (including safety lab parameters).

Secondary Endpoints:

1. Improvement in the scoring of breath holds and hyperventilation, as measured with non-invasive respiratory inductance plethysmography (NoxT3 device) and parents' diaries.
2. Changes in general behaviour, communication, feeding and motor skills as assessed by the investigator (based on Kerr and Naidu validated severity scores) and recorded in parents' diary.
3. Decrease in seizure frequency as reported in parents' diary.
4. Improvement in sleep schedule as recorded in a sleep diary.
5. Change in height and weight. Population:Ten girls, 6 to 15 years old, diagnosed with Rett syndrome (RTT) Study Design:This is a single - center, exploratory, open-label, study in 10 girls diagnosed with RTT. The study will consist of four parts: Screening and baseline assessments, initial and final dose-setting period, treatment period and end-of study follow-up.

Investigational Product:Glatiramer Acetate (Copaxone® , Teva Pharmaceutical Industries Ltd.) Sample Size Consideration: The planned sample size of 10 patients was considered adequate by the investigator for this phase I exploratory proof-of-concept study. The study is not expected to show statistical significance or statistical power, only a trend for the study endpoints. Each patient will serve as her own control.

Duration of Study: Approximately 8 months per patient (including up to 2 weeks pre-treatment assessment, 6 months initial dose and treatment periods and end-of study visit).

Overall study duration: the study is expected to be completed within 12 months (dependent on rate of recruitment).

ELIGIBILITY:
Inclusion Criteria:

1. Females, age 6-15 years (inclusive).
2. Patients whose parents or legal custodians have provided written informed consent to participate in the study.
3. A diagnosis of RTT (classical or variant), defined according to the internationally agreed 2010 RetSearch criteria [4].
4. Evidence of a genetically defined pathological change in the MECP2 gene (point mutation or deletion)
5. Patients with known epileptiform activity as recorded on EEG.
6. Blood pressure and heart rate within normal limits (blood pressure: systolic 90-140 mmHg; diastolic 50-90 mmHg, heart rate 40-120 beats per minute
7. An electrocardiogram (ECG) which, according to the Investigator's judgment does not contraindicate participation in the study.
8. No clinically significant abnormalities in haematology, blood chemistry lab tests at screening.
9. Parents must be able to understand the requirements of the study and must be willing to comply with the requirements of the study

Exclusion Criteria:

1. Any medical problem or chronic illness beyond those known to be associated with Rett Syndrome which, in the investigator's judgment, contraindicates administration of the study medication.
2. Severe respiratory dysfunction (defined as tracheostomy and/or chronic oxygen therapy at least 4 hours a day and/or repeated aspiration pneumonia - at least 4 in the last year).
3. Intractable seizures that started during the last 6 months prior to beginning of the study.
4. Known hypersensitivity to glatiramer or mannitol.
5. Participation in another clinical study.
6. Parents of a patient who are unable to communicate well with the investigator and staff and comply with study procedures and follow-up
7. Parents of a patient who are unwilling to sign consent form.

Ages: 6 Years to 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-09 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Improvement of epileptiform activity as recorded in a 24-hours EEG. | 6 months

SECONDARY OUTCOMES:
1.Improvement in the scoring of breath holds and hyperventilation, as measured with non-invasive respiratory inductance plethysmography (NoxT3 device) and parents' diaries. | 8 months
2. Changes in general behaviour, communication, feeding and motor skills as assessed by the investigator (based on Kerr and Naidu validated severity scores) and recorded in parents' diary. | 8 months
Decrease in seizure frequency as reported in parents' diary. | 8 months
Improvement in sleep schedule as recorded in a sleep diary. | 8 months
Change in height and weight | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Bruria Ben Zeev, prof., Principal Investigator — Sheba Medical Center; Andreea Nissenkorn, Dr., Principal Investigator — Sheba Medical Center; Irit Avisar, R.N M.A, Study Director — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel